CLINICAL TRIAL: NCT01706224
Title: Sero-prevalence of Pertussis Antibodies and Disease Awareness Among Healthcare Professionals in Spain
Brief Title: Sero-prevalence of Anti-pertussis Antibodies and Disease Awareness Among Spanish Healthcare Professionals
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 115539
Record Dates: First submitted 2012-09-27; First posted 2012-10-15 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Pertussis
Keywords: Pertussis antibodies; Bordetella pertussis; sero-prevalence; Healthcare professionals (HCP); Spain
MeSH Terms: conditions — Whooping Cough | interventions — Blood Specimen Collection; Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood

GROUPS / COHORTS (4):
- Group A: Subjects in this group will be all physicians actively working at hospital centres in Spain.
  Interventions: Procedure: Blood sample; Other: Data collection
- Group B: Subjects in this group will be all nurses actively working at hospital centres in Spain.
  Interventions: Procedure: Blood sample; Other: Data collection
- Group C: Subjects in this group will be all ancillary nursing professionals actively working at hospital centres in Spain.
  Interventions: Procedure: Blood sample; Other: Data collection
- Group D: Subjects in this group will be all midwives actively working at hospital centres in Spain.
  Interventions: Procedure: Blood sample; Other: Data collection

INTERVENTIONS:
Procedure: Blood sample — Samples will be tested to determine the presence of anti-pertussis antibodies.
Other: Data collection — Electronic Case Report Forms (eCRF)
Other: Data collection — Questionnaires, active questioning.

SUMMARY:
This study aims to determine the sero-prevalence of anti-pertussis antibodies among healthcare professionals at hospital centres in Spain.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the subject.
* Subjects who the investigator believes that they can and will comply with the requirements of the protocol.
* Male and female healthcare professionals aged ≥18 years from selected hospitals.
* Healthcare professionals in frequent contact with patients in the hospitals.
* Agreeing for collection of a blood sample for the study.

Exclusion Criteria:

• Medical students working as healthcare professionals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthcare professionals actively working and involved with patient care in Spanish hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 757 (Actual)
Dates: Start 2012-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of the overall sero-prevalence of Bordetella pertussis infection among subjects with respect to anti-pertussis (anti-PT) antibody levels. | Day 0 of each subject at the time of enrollment.
Evaluation of the overall sero-prevalence of Bordetella pertussis infection among subjects with respect to anti-PT seropositivity status. | Day 0 of each subject at the time of enrollment.
Evaluation of the overall sero-prevalence of Bordetella pertussis infection among subjects with respect to anti-PT seronegativity status. | Day 0 of each subject at the time of enrollment.

SECONDARY OUTCOMES:
Evaluation of the sero-prevalence of B. pertussis antibodies among healthcare professionals aged ≥ 18 years. | Day 0 of each subject at the time of enrollment.
  By age and gender, by type of healthcare professional, by hospital department of the healthcare professional, duration of service and time spent with patients.
Evaluation of the sero-prevalence of anti-pertussis antibodies among healthcare professionals by vaccination history. | Day 0 of each subject at the time of enrollment.
Evaluation of the sero-prevalence of anti-pertussis antibodies among healthcare professionals by previous history of pertussis. | Day 0 of each subject at the time of enrollment.
Description of the knowledge and beliefs about whooping cough and vaccination against pertussis among healthcare professionals. | Day 0 of each subject at the time of enrollment.
Description of the household composition of healthcare professionals to identify the proportion of healthcare professionals potentially at a higher risk of contracting and transmitting pertussis. | Day 0 of each subject at the time of enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Spain (3):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, L'Hospitalet de Llobregat
  - GSK Investigational Site, Majadahonda

REFERENCES:
- [Derived] Rodriguez de la Pinta ML, Castro Lareo MI, Ramon Torrell JM, Garcia de Lomas J, Devadiga R, Reyes J, McCoig C, Tafalla M, Garcia-Corbeira P. Seroprevalence of pertussis amongst healthcare professionals in Spain. Vaccine. 2016 Feb 17;34(8):1109-14. doi: 10.1016/j.vaccine.2015.12.036. Epub 2015 Dec 22. PMID 26718690